CLINICAL TRIAL: NCT03001284
Title: Multiple Sclerosis Produces Cardiovascular Subclinical Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Raluca Mincu, Dr, Carol Davila University of Medicine and Pharmacy
Other Study IDs: UMFCD-141531-RM
Record Dates: First submitted 2016-12-08; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple sclerosis patients: patients with confirmed multiple sclerosis, diagnosed according to the revised McDonald's criteria
  Interventions: Other: NO intervention
- Control subjects: control subjects, matched for age, gender, and presence of cardiovascular risk factors
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention

SUMMARY:
Multiple sclerosis (MS), debilitating disease involving primarily the central nervous system, may cause cardiovascular dysfunction, due to autonomous nervous system dysfunction, physical invalidity, increased oxidative stress, and systemic inflammatory status, but the detailed mechanisms are not elucidated. The investigators aimed to assess left and right ventricular (LV and RV) function, left atrial (LA) function, arterial function, and atrial-ventricular-arterial coupling in patients with MS, compared to control subjects. LV systolic and diastolic function and RV function were assessed by 2D- and 3D- echocardiography, tissue Doppler, and speckle tracking echocardiography. LA function was assessed by LA volume index and LA strain. Arterial remodeling and stiffness were assessed by intima media-thickness, pulse wave velocity, and parameters of wave intensity and endothelial function

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;
2. patients with confirmed MS diagnosis, both newly diagnosed or already under immunomodulatory treatment;
3. informed consent signed.

Exclusion Criteria:

1. MS treated with mitoxantrone;
2. patients with known cardiovascular disease;
3. presence of other neurological conditions;
4. any renal, pulmonary, hepatic or hematological disease;
5. diabetes mellitus;
6. any degree of arterial hypertension;
7. pregnancy;
8. and difficult acoustic window

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: te investigators enrolled prospectively patients with confirmed multiple sclerosis, diagnosed according to the revised McDonald's criteria[8], and control subjects, matched for age, gender, and presence of cardiovascular risk factors.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricle systolic dysfunction - by echocardiography | 1 year
Right ventricle systolic dysfunction- by echocardiography | 1 year
Left ventricular diastolic function - by echocardiography | 1 year
arterial function - by vascular echography | 1 year

IPD SHARING:
Plan to Share IPD: No